CLINICAL TRIAL: NCT00005867
Title: Phase III Trial Comparing CHOP ot PMitCEBO in Good Risk Patients With Histologically Aggresive Non Hodgkin's Lymphoma
Brief Title: Combination Chemotherapy in Treating Patients With Aggressive Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lymphoma Trials Office (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: BNLI-CHOPVPMITCEBO-GOODRISK; CDR0000067900 (Registry Identifier: PDQ (Physician Data Query)); EU-99052
Record Dates: First submitted 2000-06-02; First posted 2003-01-27 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2007-03

CONDITIONS: Lymphoma
Keywords: stage I grade 3 follicular lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse large cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic | interventions — Bleomycin; VAP-cyclo protocol; Cyclophosphamide; Doxorubicin; Etoposide; Mitoxantrone; Prednisolone; Vincristine

INTERVENTIONS:
Biological: bleomycin sulfate
Drug: CHOP regimen
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: mitoxantrone hydrochloride
Drug: prednisolone
Drug: vincristine sulfate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. It is not yet known which regimen of combination chemotherapy is most effective for non-Hodgkin's lymphoma.

PURPOSE: This randomized phase III trial is studying two regimens of combination chemotherapy and comparing how well they work in treating patients with aggressive non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the overall survival, failure free survival, disease specific survival, relapse free survival, and response rate in patients with aggressive non-Hodgkin's lymphoma treated with mitoxantrone, cyclophosphamide, etoposide, vincristine, bleomycin, and prednisolone (PMitCEBO) versus cyclophosphamide, doxorubicin, vincristine, and prednisolone (CHOP).
* Compare the early and late toxicities of these regimens in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to one of two treatment arms.

* Arm I: Patients receive mitoxantrone IV, cyclophosphamide IV, and etoposide IV on day 1 and vincristine and bleomycin IV on day 8. Treatment continues every 14 days for a maximum of 8 courses in the absence of disease progression or unacceptable toxicity. Patients also receive oral prednisolone daily on courses 1 and 2 and every other day beginning on course 3 and continuing until the end of treatment.
* Arm II: Patients receive cyclophosphamide IV, doxorubicin IV, and vincristine IV on day 1 and oral prednisolone on days 1-5. Treatment continues every 21 days for a maximum of 8 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed at 4 weeks, then every 3 months for 1 year, every 6 months for 5 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 310 patients (155 per arm) will be accrued for this study over 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven previously untreated bulky stage IA or stage IB-IV aggressive non-Hodgkin's lymphoma of 1 of the following types:

  * Working formulation:

    * Follicular large cell
    * Diffuse mixed cell
    * Diffuse large cell
    * Diffuse immunoblastic OR
  * REAL classification:

    * Diffuse large B-cell
    * Peripheral T-cell
* Measurable or evaluable disease
* Good prognosis defined as no more than one of the following:

  * Stage III/IV disease
  * LDH greater than upper limit of normal
  * ECOG/WHO 2-4
* No lymphoblastic or Burkitt's lymphoma
* No CNS involvement

PATIENT CHARACTERISTICS:

Age:

* 18 to 59

Performance status:

* See Disease Characteristics

Life expectancy:

* Not specified

Hematopoietic:

* Hemoglobin at least 10 g/dL
* Neutrophil count at least 2,000/mm3
* Platelet count at least 100,000/mm3

Hepatic:

* Bilirubin, AST, and ALT no greater than 1.5 times upper limit of normal

Renal:

* Creatinine no greater than 1.7 mg/dL

Cardiovascular:

* Ejection fraction at least 50% unless dysfunction attributable to lymphoma

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other concurrent serious uncontrolled medical conditions
* No other prior malignancy except adequately treated nonmelanoma skin cancer or cervical intraepithelial neoplasia

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy to more than 35% of hematopoietic sites
* Concurrent consolidation radiotherapy allowed

Surgery:

* Not specified

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 310 (Estimated)
Dates: Start 1998-01; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Overall survival in patients treated with mitoxantrone, cyclophosphamide, etoposide, vincristine, bleomycin, and prednisolone (PMitCEBO) versus cyclophosphamide, doxorubicin, vincristine, and prednisolone (CHOP)

SECONDARY OUTCOMES:
Failure-free survival, disease specific survival, relapse-free survival, death due to toxicity, response rate, and toxicity at 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Pettengell, MD, Study Chair — St. George's Hospital
Locations (46):
- United Kingdom (46):
  - Stoke Mandeville Hospital, Aylesbury-Buckinghamshire, England
  - Horton Hospital, Banbury, England
  - Basildon University Hospital, Basildon, England
  - Birmingham Heartlands Hospital, Birmingham, England
  - Bradford Hospitals NHS Trust, Bradford, England
  - Bristol Haematology and Oncology Centre, Bristol, England
  - Addenbrooke's Hospital at Cambridge University Hospitals NHS Foundation Trust, Cambridge, England
  - Cheltenham General Hospital, Cheltenham, England
  - Countess of Chester Hospital NHS Foundation Trust, Chester, England
  - Saint Richards Hospital, Chichester, England
  - Essex County Hospital, Colchester, England
  - Walsgrave Hospital, Coventry, England
  - Russells Hall Hospital, Dudley, England
  - Chase Farm Hospital, Enfield, England
  - Medway Maritime Hospital, Gillingham Kent, England
  - Hull Royal Infirmary, Hull, England
  - Hinchingbrooke Hospital, Huntingdon, England
  - Queen Elizabeth Hospital, Kings Lynn, England
  - Leicester Royal Infirmary, Leicester, England
  - Royal Liverpool and Broadgreen Hospitals NHS Trust, Liverpool, England
  - Aintree University Hospital, Liverpool, England
  - Saint Bartholomew's Hospital, London, England
  - St. Thomas' Hospital, London, England
  - St. George's Hospital, London, England
  - Middlesex Hospital, London, England
  - Clatterbridge Centre for Oncology NHS Trust, Merseyside, England
  - Norfolk and Norwich University Hospital, Norwich, England
  - Nottingham City Hospital NHS Trust, Nottingham, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Pontefract General Infirmary, Pontefract West Yorkshire, England
  - Oldchurch Hospital, Romford, England
  - Scunthorpe General Hospital, Scunthorpe, England
  - Cancer Research Centre at Weston Park Hospital, Sheffield, England
  - Southampton University Hospital NHS Trust, Southampton, England
  - University Hospital of North Staffordshire, Stoke-On-Trent Staffs, England
  - East Surrey Hospital, Surrey, England
  - Royal Marsden NHS Foundation Trust - Surrey, Sutton, England
  - Sandwell General Hospital, West Bromwich, England
  - Cancer Care Centre at York Hospital, York, England
  - Centre for Cancer Research and Cell Biology at Belfast City Hospital, Belfast, Northern Ireland
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Pinderfields Hospital NHS Trust, Wakefield, Scotland
  - Ysbyty Gwynedd, Bangor, Wales
  - University Hospital of Wales, Cardiff, Wales
  - Glan Clywd District General Hospital, Rhyl, Denbighshire, Wales
  - Mount Vernon Cancer Centre at Mount Vernon Hospital, Rhyl, Denbighshire, Wales